CLINICAL TRIAL: NCT00606632
Title: A Comparative Study of PET/CT Versus Diagnostic CT for the Detection of Clear Cell Renal Cell Carcinoma in Pre-surgical Patients With Renal Masses Using Iodine-124 Labeled Chimeric G250 (124I-cG250)
Brief Title: Pre-surgical Detection of Clear Cell Renal Cell Carcinoma (ccRCC) Using Radiolabeled G250-Antibody
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WX/20-001
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
Keywords: Renal Mass; Clear Cell Renal Cell Carcinoma; Cancer of Kidney; Kidney Cancer; Neoplasms; cG250; antibody, monoclonal; Iodine 124; Positron-Emission Tomography; Kidney; Renal Cancer; Renal Neoplasms
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 124-Iodine-cG250 (124I-cG250) (Other): Single arm study, comparing 124I cG250 PET/CT and CT. Each patient underwent a PET/CT and CT scan days (+/-2days) after receipt of 124I cG250.
  Interventions: Drug: 124-Iodine-cG250 (124I-cG250); Procedure: CT

INTERVENTIONS:
Drug: 124-Iodine-cG250 (124I-cG250) — i.v. and PET/CT scan 4+/-2 days after administration
  Other Names: Ca9-SCAN
Procedure: CT — contrast enhanced CT scan

SUMMARY:
This is a multicenter Phase III study to demonstrate the diagnostic utility of 124I-cG250 PET/CT pre-surgical imaging in patients with operable renal masses.

DETAILED DESCRIPTION:
A preoperative 124I-cG250 PET scan may distinguish between clear cell and non-clear cell renal carcinoma in patients with renal masses. Studies of imaging characteristics of 124I by a variety of PET cameras, quantification of tumor uptake of 124I-labeled antibody and correlation with biopsy measurement of tumor and normal tissue have met with encouraging results. As clear cell renal cancers are associated with an aggressive phenotype their a priori determination may help guide appropriate surgical/therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Subject is over 18 years of age.
* Presence of a renal mass.
* Scheduled for surgical resection of renal mass (partial or total nephrectomy, open or laparoscopic technique).
* Expected survival of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2.
* The following laboratory results should be within the following limits within the last 2 weeks prior to study day 1:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Serum bilirubin ≤ 2.0 mg/dL
  * Aspartate aminotransaminase (AST) ≤ 2.5 x ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Serum creatinine ≤ 2.0 mg/dL (calculated creatinine clearance >45 ml/min)
* Negative serum pregnancy test; to be performed on female patients of childbearing potential within 24 hours prior to receiving investigational product. All females of childbearing potential must indicate intent to avoid pregnancy and must use an accepted, effective method of contraception for the duration of the study.
* Recovered from toxicity of any prior therapy.
* Able and willing to give valid written informed consent.

Exclusion Criteria:

* Metastasis of primary tumor other than Renal Cell Carcinoma (RCC).
* Prior history of malignancy within the last 5 years.
* Prior exposure to murine proteins or chimeric antibodies.
* Intercurrent medical condition that may limit the amount of antibody to be administered.
* Intercurrent medical condition that renders the patient ineligible for surgery.
* New York Heart Association Class III/IV cardiac disease.
* History of autoimmune hepatitis.
* Chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to 124I-cG250 infusion on day 1.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Lack of availability for immunological and clinical follow-up assessments.
* Participation in any other clinical trial involving another investigational product within 4 weeks prior to enrolment.
* Women who are pregnant or breastfeeding.
* Allergy to iodine, hyperthyroidism, or Grave's Disease.
* Known allergic reaction to human serum albumin.
* Contraindication for contrast-enhanced CT or PET/CT.
* Contraindication to potassium iodide intake (see package insert).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2008-03; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaitanya Divgi, MD, Principal Investigator — University of Pennsylvania
Locations (14):
- United States (14):
  - David Geffen School of Medicine, UCLA, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - H. Lee Moffitt Cancer Center & Research Center, Tampa, Florida
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UNC School of Medicine-Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas

REFERENCES:
- [Background] Divgi CR, Pandit-Taskar N, Jungbluth AA, Reuter VE, Gonen M, Ruan S, Pierre C, Nagel A, Pryma DA, Humm J, Larson SM, Old LJ, Russo P. Preoperative characterisation of clear-cell renal carcinoma using iodine-124-labelled antibody chimeric G250 (124I-cG250) and PET in patients with renal masses: a phase I trial. Lancet Oncol. 2007 Apr;8(4):304-10. doi: 10.1016/S1470-2045(07)70044-X. PMID 17395103
- [Derived] Divgi CR, Uzzo RG, Gatsonis C, Bartz R, Treutner S, Yu JQ, Chen D, Carrasquillo JA, Larson S, Bevan P, Russo P. Positron emission tomography/computed tomography identification of clear cell renal cell carcinoma: results from the REDECT trial. J Clin Oncol. 2013 Jan 10;31(2):187-94. doi: 10.1200/JCO.2011.41.2445. Epub 2012 Dec 3. PMID 23213092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 226 subjects were enrolled at 14 study sites in the USA.
Groups:
- PET/CT Versus CT: PET/CT and CT scans for all study subjects 4 days (+/- 2 days) after 124I cG250 administration.
Period: Overall Study
Arm/Group | PET/CT Versus CT
Started | 226
Completed | 204
Not Completed | 22
Not completed — Withdrawal by Subject | 13
Not completed — Miscellaneous reasons | 9

BASELINE CHARACTERISTICS:
Groups:
- PET/CT Versus CT: All subjects were scheduled to receive a PET/CT and a diagnostic CT
Arm/Group | PET/CT Versus CT
Number analyzed (Participants) | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 167
  >=65 years | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 142
Region of Enrollment [Number; unit: participants]
  United States | 226

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of 124I-cG250 PET/CT Versus Diagnostic CT.
Description: Average estimate of three independent, blinded central readers per imaging modality on the proportion of participants that were correctly identified on the 124I-cG250 PET/CT Images of having (sensitivity) or not having (specificity) clear cell renal carcinoma (ccRCC) compared to CT images.
  Histopathology provided the standard-of-truth because it is the only definitive method for accurately identifying ccRCC.
Time Frame: 6 months
Population: ITD (Intend-to-Diagnose) observed case: All subjects who were enrolled and infused with the investigational product and who had a "standard-of-truth" (histopathology) result and images evaluated as readable by the blinded readers
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Groups:
- Sensitivity CT: Sensitivity of diagnostic CT scan for proportion of patients with positive histology (ccRCC) and evaluable images.
  The sensitivity refers to the ability of the diagnostic test to correctly identify those patients with the disease, in this case ccRCC.
- Sensitivity PET/CT: Sensitivity of 124I-cG250 PET/CT scan for proportion of patients with positive histology (ccRCC) and evaluable images.
  The sensitivity refers to the ability of the diagnostic test to correctly identify those patients with the disease, in this case ccRCC.
- Specificity PET/CT: Specificity of 124I-cG250 PET/CT scan for proportion of patients with negative histology (no ccRCC) and evaluable images.
  The specificity of refers to the ability of the diagnostic test to correctly identify those patients without the disease (in this case non-ccRCC).
- Specificity CT: Specificity of CT scan for proportion of patients with negative histology (no ccRCC) and evaluable images.
  The specificity refers to the ability of the diagnostic test to correctly identify those patients without the disease (in this case non-ccRCC).
Arm/Group | Sensitivity CT | Sensitivity PET/CT | Specificity PET/CT | Specificity CT
Number analyzed (Participants) | 143 | 143 | 52 | 52
Proportion of participants | 0.76 [0.63 to 0.88] | 0.86 [0.75 to 0.97] | 0.86 [0.69 to 1.0] | 0.47 [0.19 to 0.75]
Statistical Analysis 1: Comparison: Sensitivity CT vs Sensitivity PET/CT; Test type: Superiority; p = 0.023, McNemar
Statistical Analysis 2: Comparison: Specificity PET/CT vs Specificity CT; Test type: Superiority; p < 0.01, McNemar

2. Secondary Outcome: Accuracy of 124I-cG250 PET/CT Imaging Versus Diagnostic CT Imaging
Description: The Accuracy is the proportion of participants with correct determinations of 124I-cG250 PET/CT imaging compared to diagnostic CT Imaging in the detection of ccRCC as confirmed by histopathology diagnoses. The numbers represent the average estimate of three independent, blinded central readers per imaging modality. For the secondary efficacy variables no 95% CIs for differences of averages were calculated.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Groups:
- PET/CT: Patients with 124I-cG250 PET/CT evaluable images.
- Diagnostic CT: Patients with diagnostic CT images.
Arm/Group | PET/CT | Diagnostic CT
Number analyzed (Participants) | 195 | 195
Proportion of participants | 0.86 | 0.68

3. Secondary Outcome: Positive Predictive Value (PPV)
Description: The Positive Predictive Value (PPV) reflects the Proportion of positive results that are true positive. The PPV of 124I-cG250 PET/CT imaging compared to diagnostic CT Imaging in the detection of ccRCC as confirmed by histopathology diagnoses. The numbers represent the average estimate of three independent, blinded central readers per imaging modality. For the secondary efficacy variables no 95% CIs for differences of averages were calculated.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Protportion of participants
Arm/Group | PET/CT | Diagnostic CT
Number analyzed (Participants) | 195 | 195
Protportion of participants | 0.94 | 0.80

4. Secondary Outcome: Negative Predictive Value (NPV)
Description: Negative Predictive Value (NPV) reflects the proportion of negative results that are true negatives. The NPV of 124I-cG250 PET/CT imaging compared to diagnostic CT Imaging in the detection of ccRCC as confirmed by histopathology diagnoses. The numbers represent the average estimate of three independent, blinded central readers per imaging modality. For the secondary efficacy variables no 95% CIs for differences of averages were calculated.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | PET/CT | Diagnostic CT
Number analyzed (Participants) | 195 | 195
Proportion of participants | 0.69 | 0.41

ADVERSE EVENTS:
Arm/Group | PET/CT Versus CT
Serious Adverse Events (participants affected / at risk) | 33/226
Other Adverse Events (participants affected / at risk) | 191/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET/CT Versus CT (N=226)
Nausea (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Disease Progression (General disorders) | 1 (1)
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Extravasation of urine (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinoma (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET/CT Versus CT (N=226)
Procedural pain (Injury, poisoning and procedural complications) | 27 (27)
Nausea (Gastrointestinal disorders) | 44 (44)
Constipation (Gastrointestinal disorders) | 26 (26)
Fatigue (General disorders) | 26 (26)
Abdominal pain (Gastrointestinal disorders) | 25 (25)
Headache (Nervous system disorders) | 24 (24)
Diarrhoea (Gastrointestinal disorders) | 19 (19)
Incision site pain (Injury, poisoning and procedural complications) | 19 (19)
Insomnia (Psychiatric disorders) | 19 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15)
Anxiety (Psychiatric disorders) | 14 (14)
Dizziness (Nervous system disorders) | 14 (14)
Vomitting (Gastrointestinal disorders) | 13 (13)
Dysgeusia (Nervous system disorders) | 12 (12)
Pain (General disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less